CLINICAL TRIAL: NCT05209984
Title: A Phase 3, Randomized, Double-blind, Double-dummy, Parallel-group, Active Drug and Placebo-controlled, Safety, Efficacy and Superiority of Sibutramine IR/Topiramate XR in Overweight Adults With Comorbidities/Obesity
Brief Title: A Phase 3, Double-blind/Double-dummy, Safety/Efficacy/Superiority of Sibutramine/Topiramate XR in Adults With Overweight
Acronym: UNLIMITED
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic change in development priorities
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF178
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — sibutramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental drug (Sibutramine IR 15mg / Topiramate XR 75mg) (Experimental): ADF1 Group Eurofarma drug association of sibutramine IR 15mg / topiramate XR 75mg
  Interventions: Drug: ADF1 Group Eurofarma drug association of Sibutramine IR 15mg / Topiramate XR 75mg
- Experimental drug (Sibutramine IR 15mg / Topiramate XR 100mg) (Experimental): ADF2 Group Eurofarma drug association of sibutramine IR 15mg (Sibus®) Topiramate XR 100mg from Eurofarma Laboratórios S.A..
  Interventions: Drug: ADF2 Group Eurofarma drug association of Sibutramine IR 15mg / Topiramate XR 100mg
- Sibus (Sibutramine 15mg) (Active Comparator): SIB Group Sibutramine 15mg
  Interventions: Drug: SIB Group Sibus (Sibutramine) 15mg
- Placebo Group (Placebo Comparator): Placebo Group
  Interventions: Drug: Placebo Group

INTERVENTIONS:
Drug: ADF1 Group Eurofarma drug association of Sibutramine IR 15mg / Topiramate XR 75mg — Participant will receive for two (2) weeks one (01) ADF sibutramine IR/topiramate XR 5mg/25mg placebo capsule once daily + one (01) sibutramine placebo capsule 10mg; after that 2 weeks, participants will receive one (01) placebo capsule of ADF sibutramine IR/ topiramate XR 5mg/25mg once daily + one (01) capsule of ADF sibutramine IR/ topiramate XR 5mg/25mg once daily + one (01) 10mg sibutramine placebo capsule; after this period, they will receive two (02) capsules of ADF sibutramine IR/topiramate XR 5mg/25mg (totaling 10mg of sibutramine and 50mg of topiramate) + a placebo capsule of ADF sibutramine IR/topiramate XR 5mg/25mg once a day + one (one) 10mg sibutramine placebo capsule, taken once daily, for two (02) additional weeks, on the titration scheme. On the treatment period, will receive one (01) ADF Sibutramine IR/Topiramate XR 15mg/75mg capsule + one (01) Sibutramine IR 15mg placebo capsule (Sibus®) + one (01) Topiramate XR 100mg placebo capsule, once daily, for 52 weeks.
  Other Names: EF178 15/75mg
  Arms: Experimental drug (Sibutramine IR 15mg / Topiramate XR 75mg)
Drug: ADF2 Group Eurofarma drug association of Sibutramine IR 15mg / Topiramate XR 100mg — Participant will receive for two (02) weeks one (01) capsule of ADF sibutramine IR/topiramate XR 5mg/25mg once daily + one (01) capsule of placebo sibutramine 10mg; after this initial period of 2 weeks, participants will receive (02) ADF sibutramine IR/topiramate XR 5mg/25mg capsules (totaling 10mg of sibutramine and 50mg of topiramate) + one (01) 10mg sibutramine placebo capsule, taken once daily, for two (02) weeks; after this period, they will receive three (03) capsules of ADF sibutramine IR/topiramate XR 5mg/25mg (totaling 15mg of sibutramine and 75mg of topiramate) + one (01) capsule of 10mg sibutramine placebo, taken once daily, for two ( 02) additional weeks, on titration scheme. On the treatment period, will receive one (01) Sibutramine IR 15mg capsule (Sibus®) + one (01) Topiramate XR 100mg capsule + one (01) ADF placebo capsule sibutramine IR/topiramate XR 15mg/75mg, taken once daily, taken once daily, for 52 weeks.
  Other Names: EF178 15/100mg
  Arms: Experimental drug (Sibutramine IR 15mg / Topiramate XR 100mg)
Drug: SIB Group Sibus (Sibutramine) 15mg — Participant will receive for two (02) weeks one (01) 10mg sibutramine placebo capsule + one (01) 5mg/25mg sibutramine ADF placebo capsule IR/topiramate XR; after this initial period, they will receive for two (02) weeks one (01) 10mg sibutramine capsule + two (02) placebo capsules of ADF sibutramine IR/topiramate XR 5mg/25mg; after this 4-week period, participants will receive one (01) 10mg sibutramine capsule and three (03) ADF sibutramine IR/topiramate XR 5mg/25mg placebo capsules, taken once daily, for two (02) additional weeks. This corresponds to the titration scheme.On the treatment period, patient will receive one (01) Sibutramine 15mg capsule + one (01) Sibutramine IR/topiramate XR 15mg/75mg placebo capsule + one (01) placebo capsule of Topiramate XR 100mg, taken once daily, for 52 weeks.
  Other Names: Sibutramine 15mg
  Arms: Sibus (Sibutramine 15mg)
Drug: Placebo Group — participants randomized to the Placebo Group will receive for two (02) weeks one (01) 10mg sibutramine placebo capsule + one (01) sibutramine IR/ topiramate XR 5mg/25mg placebo capsule; after this initial period, they will receive one (01) sibutramine 10mg placebo capsule + two (02) sibutramine IR/ topiramate XR 5mg/25mg placebo capsules, taken once daily, for two (02) weeks; after this 4-week period, participants will receive one (01) 10mg sibutramine placebo capsule + three (03) ADF placebo capsules, taken once daily, for two (02) weeks.On the treatment period, patient will receive one (01) Sibutramine 15mg placebo capsule + one (01) ADF sibutramine IR/Topiramate XR 15mg/75mg placebo capsule + one (01) Topiramate XR 100mg placebo capsule, in once daily intake for 52 weeks.
  Other Names: Ef178 Placebo
  Arms: Placebo Group

SUMMARY:
A phase 3, multicenter, randomized, double-blind, double-dummy, parallel-group, active-drug- and placebo-controlled clinical trial to assess the safety, efficacy and superiority of the new fixed-dose combination sibutramine IR/topyramat XR in weight reduction in overweight adults with comorbidity(ies) or obesity

DETAILED DESCRIPTION:
A phase 3, multicenter, national, randomized, double-blind, double-dummy, parallel-group, active-drug and placebo-controlled, superiority clinical trial. Individuals of both sexes aged ≥18 years and ≤60 years, overweight (BMI ≥ 27kg/m2) in the presence of comorbidities (dyslipidemia, systemic arterial hypertension [SAH], pre-diabetes and/or sleep apnea) or obese (BMI ≥ 30kg/m2 and < 45kg/m2).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged between 18 and 60 years (inclusive);
2. BMI ≥ 27kg/m2 and < 45kg/m2. Patients with a BMI ≥ 27kg/m2 and < 30kg/m2 must have at least one of the following comorbidities to be included in the study: dyslipidemia, systemic arterial hypertension (SAH), pre-diabetes (fasting glucose ≥ 100mg/dL and < 126 mg/dL and/or HbA1c ≥ 5.7% and < 6.5%] and/or sleep apnea (confirmed by polysomnography performed up to three months before enrollment in the study);
3. Women of childbearing age must use adequate contraceptive methods;
4. Volunteers willing and able to comply with all aspects of the protocol;
5. Signing the Informed Consent Form (ICF) before performing any study procedure.

Exclusion Criteria:

1. Participation in a lifestyle change program within the three months prior to the start of the study;
2. Treatment with drugs (prescription or over-the-counter) or alternative drugs intended to promote weight loss within the three months prior to the start of the study. These medications include, among others: liraglutide, orlistat, sibutramine, topiramate, naltrexone, bupropion, sertraline, fluoxetine, duloxetine. Note: The use of metformin or other hypoglycemic drugs prescribed for the treatment of polycystic ovary syndrome or prevention of diabetes is not permitted;
3. Treatment with drugs known to cause significant weight gain within three months of starting the study. These medications include, among others: corticosteroids, tricyclic antidepressants, atypical antipsychotics, and mood stabilizers (such as imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid and its derivatives, lithium).
4. Presence of diabetes mellitus;
5. History of coronary artery disease (angina, history of myocardial infarction);
6. Congestive heart failure;
7. History of tachycardia;
8. History of peripheral obstructive arterial disease;
9. History of arrhythmia;
10. History of cerebrovascular disease (stroke or transient ischemic attack);
11. Inadequately controlled systemic arterial hypertension (> 145/90 mmHg);
12. History or active pulmonary arterial hypertension;
13. History or presence of eating disorders such as bulimia and anorexia;
14. Moderate or severe renal impairment (estimated creatinine clearance < 70 mL/min);
15. Hepatic failure Child-Pugh categories B or C (Child-Pugh scale score ≥ 7 points);
16. Current use of monoamine oxidase inhibitors (MAOIs) or any other drug treatment for psychiatric disorders;
17. History of psychiatric disorder requiring previous drug treatment;
18. Glaucoma or high intraocular pressure;
19. Unstable thyroid disease or replacement therapy;
20. Hypersensitivity to sibutramine, topiramate, or to any component of the investigational product formulation;
21. Known hypersensitivity to any component of the investigational drug formulation;
22. Urinary lithiasis;
23. Pregnancy or lactation;
24. Any medical or other condition that, in the opinion of the investigator(s), prevents the participant from participating in the clinical trial, such as significantly abnormal laboratory results or any physical or mental condition that prevents compliance with the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 58 weeks
  The difference in mean percent body weight loss between the ADF sibutramine IR/topiramate XR group and the placebo-treated group is ≥5% in favor of ADF.
The mean percentage loss of body weight | 58 weeks
  The mean percentage loss of body weight in the ADF sibutramine IR/topiramate XR group was greater than that observed in the group treated with sibutramine IR

SECONDARY OUTCOMES:
Proportion of participants with weight reduction ≥ 5% | 58 weeks
  Proportion of participants with weight reduction ≥ 5% at the end of treatment in relation to baseline weight;
Proportion of participants with weight reduction ≥ 10% | 58 weeks
  Proportion of participants with weight reduction ≥ 10% at the end of treatment in relation to baseline weight
Proportion of participants with weight reduction ≥ 15% | 58 weeks
  Proportion of participants with weight reduction ≥ 15% at the end of treatment in relation to baseline weight;
Abdominal circumference | 58 weeks
  The measurement of abdominal circumference

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Eurofarma Laboratórios S.A, São Paulo, São Paulo
  - HC-FMUSP, São Paulo, São Paulo